CLINICAL TRIAL: NCT07168967
Title: The Relationship Between Adherence to the EAT-Lancet Diet and Chronotype and Psychological Well-Being: A Study in Obese Individuals
Brief Title: EAT-Lancet Diet, Chronotype, and Well-Being in Obesity
Status: Completed | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Nurefşan KONYALIGİL ÖZTÜRK, Assist. Prof. Dr, Abant Izzet Baysal University
Other Study IDs: AIBU-BD-NKÖ-02
Record Dates: First submitted 2025-09-04; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Obesity
Keywords: Chronotype; Obesity; Psychological well-being
MeSH Terms: conditions — Obesity; Psychological Well-Being

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals with obesity: This cohort includes adult participants diagnosed with obesity (BMI ≥30 kg/m²). No control group is included.

SUMMARY:
The aim of this study is to examine the relationship between the Planetary Health Diet (EAT-Lancet) dietary pattern, chronotype, and psychological well-being in obese individuals. A total of 97 individuals diagnosed with obesity were included in the study. A questionnaire form containing sociodemographic characteristics was administered to volunteers who agreed to participate in the study. In addition, participants' anthropometric measurements (body weight, height, waist and hip circumference, Body Mass Index (BMI)), biochemical parameters (fasting blood glucose, HbA1c, triglycerides, LDL-cholesterol, triglycerides, total cholesterol, C-reactive protein (CRP)), and nutritional status (food consumption record and frequency) were obtained. The Morningness-Eveningness Questionnaire was used to determine chronotype. The Psychological Well-Being Scale was used for psychological assessment.

DETAILED DESCRIPTION:
Mood disorders are common in obese individuals, and anxiety and depression often contribute to weight gain through emotional eating and inactivity. Therefore, including psychological support in obesity prevention and treatment programs is important for long-term weight loss goals. However, chronotype, which describes an individual's behavioral preferences such as sleep timing and eating, is also an important factor in determining both physical and mental health outcomes. An inappropriate chronotype has been associated with a more unfavorable body composition, poor mental health, and an increased risk of depression and anxiety. A review of the literature reveals no studies that simultaneously address the Planetary Health Diet (EAT-Lancet) dietary model, chronotype, and psychological well-being variables in obese individuals; this highlights the originality and necessity of the present study. The aim of this study is to examine the relationship between the EAT-Lancet dietary model, chronotype, and psychological well-being in obese individuals.

ELIGIBILITY:
Inclusion Criteria:

* Individuals over 19 years of age
* Individuals who are literate
* Individuals diagnosed with obesity

Exclusion Criteria:

* Individuals who have had an acute infection or inflammatory disease within the past month
* Individuals with chronic infectious or inflammatory diseases
* Individuals with cancer

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study was designed as a cross-sectional study. The study was conducted on 97 individuals aged 19-64 who were diagnosed with obesity and volunteered to participate in the study at the Diet Clinic of Izzet Baysal Physical Therapy and Rehabilitation Education and Research Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Questionnaire Form | 3 months
  Sociodemographic characteristics of the individuals (age, gender, smoking and alcohol use, constipation status, swallowing-chewing problem) were questioned.
Body Weight (BW) | 3 months
  BW was measured using a calibrated digital scale placed on a flat, tiled surface. The scale was sensitive to 100 grams.
Height | 3 months
  Height was measured using a stadiometer with the participant's head positioned in the Frankfort plane and feet placed together.
Waist Circumference (WC) | 3 months
  WC was measured at the midpoint between the lowest rib and the iliac crest (cristal point) using a flexible measuring tape.
Hip Circumference (HC) | 3 months
  HC was measured at the widest point of the hips using a flexible measuring tape.
Body Mass Index (BMI) | 3 months
  BMI was calculated by dividing body weight (in kilograms) by the square of height (in meters): BMI = weight (kg) / height² (m²).
Fasting Blood Glucose | 3 months
  Fasting blood glucose was measured using standard laboratory techniques during routine outpatient visits.
Triglycerides | 3 months
  Triglyceride levels were measured via fasting blood samples analyzed in the outpatient clinic laboratory.
LDL-Cholesterol | 3 months
  LDL-cholesterol was measured from fasting serum samples using standard enzymatic colorimetric methods.
Total Cholesterol | 3 months
  Total cholesterol was measured using routine biochemical analysis in a certified laboratory.
Albumin | 3 months
  Serum albumin levels were measured using routine laboratory procedures in outpatient visits.
Vitamin D | 3 months
  Serum vitamin D (25(OH)D) levels were assessed using chemiluminescence immunoassay methods in the outpatient clinic laboratory.
Folic Acid | 3 months
  Serum folic acid levels were measured using standard automated immunoassay techniques.immunoassay methods in the outpatient clinic laboratory.
Vitamin B12 | 3 months
  Serum vitamin B12 concentrations were measured using automated chemiluminescent immunoassay.immunoassay methods in the outpatient clinic laboratory.
Food Frequency Questionnaire | 3 months
  The foods consumed by individuals in the last month were evaluated across seven different groups, including five basic food groups (meat and meat products, milk and dairy products, bread and grains, vegetables and fruits, sugar and fats), beverages, and fast food. Participants were asked how often they consumed foods and beverages in these groups; responses were collected using the following options: "every meal," "every day," "5-6 days a week," "3-4 days a week," "1-2 days a week," "once every 15 days," "once a month," and "never." To determine the average daily consumption amounts based on consumption frequency, the following coefficients were used: 3 for "every meal," 1 for "every day," 0.7855 for "5-6 times a week," 0.498 for "3-4 times a week," 0.2145 for "1-2 times a week," 0.067 for "every 15 days," and 0.033 for "once a month.
Evaluation of Food Consumption Records | 3 months
  Responses regarding food consumption frequency were calculated using food consumption frequency calculations. The amounts of food and beverages consumed were multiplied by "3" for "every meal," '1' for "every day," "0.7855" for "5-6 times a week," "0.498" for "3-4 times a week," "0.2145" for "1-2 times a week," "0.067" for "every 15 days," and "0.033" for "once a month" to obtain the average daily amounts. Energy, macronutrients, and micronutrients were calculated using the daily intake amount.
Planetary Health Diet (EAT-Lancet) | 3 months
  In this study, the EAT-Lancet diet score was used. Adherence to the EAT-Lancet diet was scored based on the estimated average daily intake of 14 dietary components. Each component was rated as 0 (non-compliance) or 1 point (compliance), resulting in a total score ranging from 0 to 14 points.
Chronotype Eating Pattern | 3 months
  Individuals' chronotype eating patterns were determined using the Morning-Evening Questionnaire. The Morning-Evening Questionnaire consists of a total of 19 questions. The questionnaire contains questions about individuals' physical and psychological performance during a 24-hour period, which time of day they perform better, and their preferences regarding sleep and wakefulness times. As a result of the evaluation, those who scored between 70 and 86 were classified as "Definitely Morning Type"; those scoring between 59 and 69 are classified as "Close to Morning Type"; those scoring between 42 and 58 are classified as "Intermediate Type"; those scoring between 31 and 41 are classified as "Close to Evening Type"; and those scoring between 16 and 30 are classified as "Definitely Evening Type."
Psychological Assessment | 3 months
  Individuals were psychologically assessed using the Psychological Well-Being Scale. The scale defines many important elements, ranging from feeling satisfied with positive relationships to having a purposeful and meaningful life. There are 8 items on the scale. Each item is answered on a scale of 1 to 7, ranging from 1 (strongly disagree) to 7 (strongly agree). When all items are answered with "strongly disagree," the total test score is 8; when answered with "strongly agree," the total test score is 56. A high score on the test indicates that the individual has abundant psychological resources and strengths.

CONTACTS AND LOCATIONS:
Overall Officials: Nurefşan Konyalıgil Öztürk, Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Bolu Abant İzzet Baysal University, Faculty of Health Sciences, Bolu, Turkey (Türkiye)